CLINICAL TRIAL: NCT00620646
Title: The Comparison of Effects Between Increased Dose of Clopidogrel and Addition of Cilostazol in Clopidogrel Non-Responders After Drug-Eluting Stent Implantation
Brief Title: The Comparison of Effects Between Increased Dose of Clopidogrel and Addition of Cilostazol
Acronym: 4C-DES
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: HC Gwon, Samsung Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2006-12-026
Record Dates: First submitted 2008-01-27; First posted 2008-02-21 (Estimated); Last update posted 2009-02-12 (Estimated); Status verified 2009-02

CONDITIONS: Clopidogrel Non-Responsiveness
Keywords: clopidogrel; platelets; percutaneous coronary intervention
MeSH Terms: interventions — Aspirin; Clopidogrel; Cilostazol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): Aspirin plus increasing clopidogrel group
  Interventions: Drug: aspirin, clopidogrel
- B (Experimental): Aspirin, clopidogrel plus cilostazol group
  Interventions: Drug: aspirin, clopidogrel, cilostazol

INTERVENTIONS:
Drug: aspirin, clopidogrel — aspirin 100 mg plus clopidogrel 150mg qd
  Arms: A
Drug: aspirin, clopidogrel, cilostazol — aspirin 100mg qd,clopidogrel 75mg qd plus cilostazol 100mg bid
  Arms: B

SUMMARY:
To compare the effect of increased dosing of clopidogrel and adding cilostazol to standard dose of clopidogrel after the insertion of drug-eluting stent in patients with clopidogrel resistance

DETAILED DESCRIPTION:
Using dual antiplatelet agents with aspirin and clopidogrel is essential after drug-eluting stent implantation to prevent restenosis and stent thrombosis. However, variable platelet response and potential resistance to therapy have emerged with clopidogrel. Several studies showed that clopidogrel resistance is associated with increased cardiovascular events after coronary interventions. New antiplatelet therapeutic strategy of is needed in case of clopidogrel resistance. We started this study to compare the effect of double dosing of clopidogrel to 150mg per day and adding cilostazol to standard dose of clopidogrel after the insertion of drug-eluting stent in patients with clopidogrel resistance.

ELIGIBILITY:
Inclusion Criteria:

* Patient with clopidogrel resistance with treatment of dual antiplatelet agent, aspirin and clopidogrel, for more than 4 weeks after drug-eluting stent
* Clopidogrel resistance is defined as a patients with platelet inhibition less than 30% in platelet function test(VerifyNow-P2Y12 assayTM, Accumetrics, San Diego, CA, USA)

Exclusion Criteria:

* Acute myocardial infarction within 2 weeks
* Unstable angina within 2 weeks
* History of using glycoprotein IIb/IIIa inhibitor within 1 month
* Cerebral infarction within 3 months
* Bleeding diathesis like coagulation disorder, thrombocytopenia (platelet count < 100,000/uL)
* history of gastrointestinal bleeding or genitourinary bleeding within 3 months
* needed oral anticoagulation
* aspirin, clopidogrel or cilostazol hypersensitivity
* congestive heart failure
* serum creatinine level >2mg/dl
* malignancy
* using cytochrome P450 inhibitor (eg, itraconazole)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2008-02; Primary Completion 2008-12 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
% platelet inhibition with VeryfyNow-P2Y12 assay, platelet function test | 4 weeks

SECONDARY OUTCOMES:
P2Y12 reaction unit (PRU) | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Hyeon-Cheol Gwon, MD, PhD, Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea